CLINICAL TRIAL: NCT07245537
Title: EndoGym Progetto di Riabilitazione Del Pavimento Pelvico e Trattamento Del Dolore Miofasciale e Dispareunia Tramite la Pratica Dello Yoga in Pazienti Con Diagnosi di Endometriosi.
Brief Title: ENDOGYM: A Holistic Approach With Pelvic Floor Physiotherapy and Yoga for Endometriosis Pain Relief
Acronym: ENDOGYM
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliero-Universitaria di Modena (Other)
Responsible Party: Principal Investigator, Carlo Alboni, MD, PhD, MD, Azienda Ospedaliero-Universitaria di Modena
Other Study IDs: 511/2024/OSS/AOUMO
Record Dates: First submitted 2025-09-29; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Endometriosis
Keywords: endometriosis; yoga; pain; quality of life; complementary therapies
MeSH Terms: conditions — Endometriosis; Pain | interventions — Yoga

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with endometriosis and chronic pelvic pain and/or dyspareunia under medical treatment: ENDOGYM consists of 12 weekly sessions over a period of 3 months. It includes two PFP sessions, lasting 1 hour each (one at the start and one at the end of the program), and 12 Yoga sessions, once a week, each lasting 60 minutes. EHP-30 questionnaire was used before and after the program to evaluate women's QoL; NRS scale was used before, half-way and after the program to evaluate CPP and dyspareunia
  Interventions: Other: Yoga; Other: Pelvic Floor Physiotherapy

INTERVENTIONS:
Other: Yoga — The Yoga sessions were designed to address specific physiological needs related to endometriosis, such as CPP, myofascial pain, chronic fatigue, and hormonal imbalance. The asanas were selected to stimulate the nervous system, promote blood circulation, and relax the pelvic muscles. The poses were adapted to avoid any direct pressure on the pelvic organs, fostering a sense of lightness and awareness. Deep breathing techniques were taught to reduce stress and improve tissue oxygenation, with a positive impact on pain management and immune function. The breathing exercises were often hypopressive to reduce the load on the pelvic area. The use of mindfulness was encouraged to increase awareness of bodily sensations, reduce anxiety, and improve emotional balance. The practice was not just "a physical activity" but an opportunity for the participant to deeply connect with her body, promoting an overall improvement in the QoL.
Other: Pelvic Floor Physiotherapy — During the two one-hour sessions of PFP, various tools were used, such as balls of different textures and a cylindrical cushion provide tactile biofeedback and help identify the boundaries of the perineum. Patients were free to adjust the intensity of the feedback by choosing or removing the appropriate aid. By perceiving the different muscular layers of the perineum and altering the posture of the pelvis and lower limbs, patients learned about perineal movements, muscle activation, and myofascial tensions. The goal was to internalize the therapeutic exercises demonstrated and apply them in various daily life situations to maintain improvements in the perineal-pelvic structures.

SUMMARY:
The aim of this study is to evaluate the combined effects of Yoga practice and pelvic floor physiotherapy (PFP) on chronic pelvic pain (CPP) and dyspareunia in endometriosis patients.

This is a retrospective study carried out from April 2024 to November 2024 conducted by University Hospital Modena (Italy). A total of 82 women with confirmed diagnosis of endometriosis were initially enrolled in the ENDOGYM program. Among them, 50 patients (61%) were therefore included in the final analysis. ENDOGYM consists of 12 weekly sessions over a period of 3 months. It includes two PFP sessions, lasting 1 hour each (one at the start and one at the end of the program), and 12 Yoga sessions, once a week, each lasting 60 minutes. EHP-30 questionnaire was used before and after the program to evaluate women's QoL; NRS scale was used before, half-way and after the program to evaluate CPP and dyspareunia.

ELIGIBILITY:
Inclusion Criteria:

* women with an ultrasound and/or post-operative histological diagnosis of endometriosis
* aged between 18-50 years
* currently undergoing medical treatment (for at least 3 months before the start of the study), and/or who have previously undergone surgical treatment
* with myofascial pain ≥ 7 (NRS scale) and deep dyspareunia ≥ 7 (NRS scale).

Exclusion Criteria:

* being pregnant
* undergoing surgery in the past 6 months
* concurrent diagnosis of fibromyalgia
* documented pelvic and/or spine trauma within 5 years of recruitment
* patients with interstitial cystitis and > 2 urinary tract infections per year, unless possibly related to endometriosis (non-bacterial)
* patients with recurrent vaginal infections, mucocutaneous inflammations of the vulva and vagina.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with an ultrasound and/or post-operative histological diagnosis of endometriosis followed at the Endometriosis and Pelvic Pain Center of the Mother-Infant Department, Institute of Obstetrics and Gynecology, University of Modena and Reggio Emilia (Italy).
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Evaluate the combined effects of Yoga practice and pelvic floor physiotherapy (PFP) on chronic pelvic pain (CPP) in endometriosis patients | From enrollment to the end of the lessons at 3 months
  Before the start of the project, a disease-specific questionnaire to measure the QoL of women with endometriosis, the Endometriosis Health Profile-30 (EHP-30) questionnaire, was used to collect data about pain, control and powerlessness, emotional well-being, social support, self-image, work life, sexual intercourse, relationship with children, the medical profession, treatment, and infertility. Response categories are evaluated using a five-point Likert scale (0-4), and each EHP-30 scale is converted into a scoring system ranging from 0 to 100, where 0 indicates the best possible health status and 100 represents the worst possible health status. The Italian version of EHP-30 was used. Finally, at the end of the project, the women completed the EHP-30 questionnaire again. Comparisons of EHP-30 total and domain scores before and after the ENDOGYM program were performed using paired t-tests (two-tailed).

SECONDARY OUTCOMES:
Evaluate the combined effects of Yoga practice and pelvic floor physiotherapy (PFP) on dyspareunia in endometriosis patients | From the enrollment till the end of the lessons at 3 months
  Before the start of the project, the NRS scale was used to collect data about deep dyspareunia in patients with endometriosis. An additional assessment of deep dyspareunia using the NRS scale was performed halfway through the process. Finally, at the end of the project, the women assessed their deep dyspareunia one last time using the NRS scale.

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Alboni, MD, Principal Investigator — AOU Policlinico di Modena
Locations (1):
- AOU Policlinico di Modena, Modena, Emilia-Romagna, Italy

REFERENCES:
- [Background] Starzec-Proserpio M, Frawley H, Bo K, Morin M. Effectiveness of nonpharmacological conservative therapies for chronic pelvic pain in women: a systematic review and meta-analysis. Am J Obstet Gynecol. 2025 Jan;232(1):42-71. doi: 10.1016/j.ajog.2024.08.006. Epub 2024 Aug 13. PMID 39142363
- [Background] Jones G, Jenkinson C, Taylor N, Mills A, Kennedy S. Measuring quality of life in women with endometriosis: tests of data quality, score reliability, response rate and scaling assumptions of the Endometriosis Health Profile Questionnaire. Hum Reprod. 2006 Oct;21(10):2686-93. doi: 10.1093/humrep/del231. Epub 2006 Jul 4. PMID 16820384
- [Background] Lee SY, Koo YJ, Lee DH. Classification of endometriosis. Yeungnam Univ J Med. 2021 Jan;38(1):10-18. doi: 10.12701/yujm.2020.00444. Epub 2020 Aug 7. PMID 32764213
- [Background] Meister MR, Sutcliffe S, Ghetti C, Chu CM, Spitznagle T, Warren DK, Lowder JL. Development of a standardized, reproducible screening examination for assessment of pelvic floor myofascial pain. Am J Obstet Gynecol. 2019 Mar;220(3):255.e1-255.e9. doi: 10.1016/j.ajog.2018.11.1106. Epub 2018 Dec 7. PMID 30527941
- [Background] Bazot M, Thomassin I, Hourani R, Cortez A, Darai E. Diagnostic accuracy of transvaginal sonography for deep pelvic endometriosis. Ultrasound Obstet Gynecol. 2004 Aug;24(2):180-5. doi: 10.1002/uog.1108. PMID 15287057
- [Background] Ravins I, Joseph G, Tene L. The Effect of Practicing "Endometriosis Yoga" on Stress and Quality of Life for Women with Endometriosis: AB Design Pilot Study. Altern Ther Health Med. 2023 Apr;29(3):8-14. PMID 35839113
- [Background] Samami E, Shahhosseini Z, Khani S, Elyasi F. Pain-focused psychological interventions in women with endometriosis: A systematic review. Neuropsychopharmacol Rep. 2023 Sep;43(3):310-319. doi: 10.1002/npr2.12348. Epub 2023 Jun 27. PMID 37366616
- [Background] Huang AJ, Rowen TS, Abercrombie P, Subak LL, Schembri M, Plaut T, Chao MT. Development and Feasibility of a Group-Based Therapeutic Yoga Program for Women with Chronic Pelvic Pain. Pain Med. 2017 Oct 1;18(10):1864-1872. doi: 10.1093/pm/pnw306. PMID 28419385
- [Background] Villemure C, Ceko M, Cotton VA, Bushnell MC. Insular cortex mediates increased pain tolerance in yoga practitioners. Cereb Cortex. 2014 Oct;24(10):2732-40. doi: 10.1093/cercor/bht124. Epub 2013 May 21. PMID 23696275
- [Background] Wojcik M, Szczepaniak R, Placek K. Physiotherapy Management in Endometriosis. Int J Environ Res Public Health. 2022 Dec 2;19(23):16148. doi: 10.3390/ijerph192316148. PMID 36498220
- [Background] van Reijn-Baggen DA, Han-Geurts IJM, Voorham-van der Zalm PJ, Pelger RCM, Hagenaars-van Miert CHAC, Laan ETM. Pelvic Floor Physical Therapy for Pelvic Floor Hypertonicity: A Systematic Review of Treatment Efficacy. Sex Med Rev. 2022 Apr;10(2):209-230. doi: 10.1016/j.sxmr.2021.03.002. Epub 2021 Jun 12. PMID 34127429
- [Background] Alboni C, Melegari S, Camacho Mattos L, Farulla A. Effects of osteopathic manipulative therapy on recurrent pelvic pain and dyspareunia in women after surgery for endometriosis: a retrospective study. Minerva Obstet Gynecol. 2024 Jun;76(3):264-271. doi: 10.23736/S2724-606X.23.05351-4. Epub 2023 Nov 23. PMID 37997320
- [Background] Del Forno S, Arena A, Pellizzone V, Lenzi J, Raimondo D, Cocchi L, Paradisi R, Youssef A, Casadio P, Seracchioli R. Assessment of levator hiatal area using 3D/4D transperineal ultrasound in women with deep infiltrating endometriosis and superficial dyspareunia treated with pelvic floor muscle physiotherapy: randomized controlled trial. Ultrasound Obstet Gynecol. 2021 May;57(5):726-732. doi: 10.1002/uog.23590. PMID 33428320
- [Background] Stratton P, Khachikyan I, Sinaii N, Ortiz R, Shah J. Association of chronic pelvic pain and endometriosis with signs of sensitization and myofascial pain. Obstet Gynecol. 2015 Mar;125(3):719-728. doi: 10.1097/AOG.0000000000000663. PMID 25730237
- [Background] Vercellini P, Somigliana E, Vigano P, Abbiati A, Daguati R, Crosignani PG. Endometriosis: current and future medical therapies. Best Pract Res Clin Obstet Gynaecol. 2008 Apr;22(2):275-306. doi: 10.1016/j.bpobgyn.2007.10.001. Epub 2007 Nov 26. PMID 18036995
- [Background] Alboni C, Cannoletta M, Mosca S, Pasini S, Farulla A, Chiossi G. Endometriosis and risk factors in pregnancy, labor and delivery: a case-control study. Minerva Obstet Gynecol. 2024 Dec;76(6):540-547. doi: 10.23736/S2724-606X.24.05527-1. Epub 2024 Nov 8. PMID 39512100
- [Background] Gambigliani Zoccoli S, La Marca A. Endometriosis affects natural and ART fertility in different ways: let's look at the whole patient and not at the single lesion. Reprod Biomed Online. 2024 Nov;49(5):104354. doi: 10.1016/j.rbmo.2024.104354. Epub 2024 Jul 3. PMID 39197400
- [Background] Barbara G, Facchin F, Buggio L, Somigliana E, Berlanda N, Kustermann A, Vercellini P. What Is Known and Unknown About the Association Between Endometriosis and Sexual Functioning: A Systematic Review of the Literature. Reprod Sci. 2017 Dec;24(12):1566-1576. doi: 10.1177/1933719117707054. Epub 2017 May 31. PMID 28558521
- [Background] Montanari G, Di Donato N, Benfenati A, Giovanardi G, Zannoni L, Vicenzi C, Solfrini S, Mignemi G, Villa G, Mabrouk M, Schioppa C, Venturoli S, Seracchioli R. Women with deep infiltrating endometriosis: sexual satisfaction, desire, orgasm, and pelvic problem interference with sex. J Sex Med. 2013 Jun;10(6):1559-66. doi: 10.1111/jsm.12133. Epub 2013 Apr 3. PMID 23551753
- [Background] Shum LK, Bedaiwy MA, Allaire C, Williams C, Noga H, Albert A, Lisonkova S, Yong PJ. Deep Dyspareunia and Sexual Quality of Life in Women With Endometriosis. Sex Med. 2018 Sep;6(3):224-233. doi: 10.1016/j.esxm.2018.04.006. Epub 2018 May 22. PMID 29801714
- [Background] Facchin F, Barbara G, Saita E, Mosconi P, Roberto A, Fedele L, Vercellini P. Impact of endometriosis on quality of life and mental health: pelvic pain makes the difference. J Psychosom Obstet Gynaecol. 2015;36(4):135-41. doi: 10.3109/0167482X.2015.1074173. Epub 2015 Aug 27. PMID 26328618
- [Background] Lemaire GS. More than just menstrual cramps: symptoms and uncertainty among women with endometriosis. J Obstet Gynecol Neonatal Nurs. 2004 Jan-Feb;33(1):71-9. doi: 10.1177/0884217503261085. PMID 14971555
- [Background] Bulletti C, Coccia ME, Battistoni S, Borini A. Endometriosis and infertility. J Assist Reprod Genet. 2010 Aug;27(8):441-7. doi: 10.1007/s10815-010-9436-1. Epub 2010 Jun 25. PMID 20574791
- [Background] Giudice LC. Clinical practice. Endometriosis. N Engl J Med. 2010 Jun 24;362(25):2389-98. doi: 10.1056/NEJMcp1000274. PMID 20573927
- [Background] Clement PB. The pathology of endometriosis: a survey of the many faces of a common disease emphasizing diagnostic pitfalls and unusual and newly appreciated aspects. Adv Anat Pathol. 2007 Jul;14(4):241-60. doi: 10.1097/PAP.0b013e3180ca7d7b. PMID 17592255